CLINICAL TRIAL: NCT03901625
Title: The Efficacy of Different Methods of Teeth Cleaning on the Levels of Volatile Sulfur Compounds in Patients With Orthodontic Fixed Appliances
Brief Title: Halitosis During Active Orthodontic Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riyadh Colleges of Dentistry and Pharmacy (Other)
Responsible Party: Principal Investigator, Omar Alkadhi, Assistant professor, Riyadh Colleges of Dentistry and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FPGRP/43734003/316
Record Dates: First submitted 2019-04-01; First posted 2019-04-03 (Actual); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Halitosis
MeSH Terms: conditions — Halitosis | interventions — Dental Devices, Home Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ManualTB+Floss (Active Comparator): Cleaning teeth with a manual toothbrush and a dental floss three times a day.
  Interventions: Device: Manual Toothbrush; Device: Dental floss
- ManualTB+Waterjet (Experimental): Cleaning teeth with a manual toothbrush and a waterjet three times a day.
  Interventions: Device: Manual Toothbrush; Device: Waterjet
- Electric TB+Floss (Experimental): Cleaning teeth with an electric toothbrush and dental floss three times a day .
  Interventions: Device: Dental floss; Device: Electric Toothbrush
- Electric TB +Waterjet (Experimental): Cleaning teeth with an electric toothbrush and a waterjet three times a day .
  Interventions: Device: Waterjet; Device: Electric Toothbrush

INTERVENTIONS:
Device: Manual Toothbrush — A manual toothbrush is used to clean teeth surfaces.
  Arms: ManualTB+Floss; ManualTB+Waterjet
Device: Dental floss — A dental floss is used to clean inter-proximal areas.
  Arms: Electric TB+Floss; ManualTB+Floss
Device: Waterjet — A waterjet is used to clean inter-proximal areas.
  Arms: Electric TB +Waterjet; ManualTB+Waterjet
Device: Electric Toothbrush — An electric toothbrush is used to clean teeth surfaces.
  Arms: Electric TB +Waterjet; Electric TB+Floss

SUMMARY:
To determine the effect of different cleaning methods and devices in reducing halitosis during active orthodontic treatment.

DETAILED DESCRIPTION:
. Observer - blind clinical trial, randomly divided into four groups, A, B, C and D. each group will undergo clinical evaluation and oral malodor assessment and they will be assigned electric or manual toothbrushes with super floss or water floss respectively.clinical evaluation will include plaque index (PI), gingival bleeding index (GBI), bracket index.and halitosis will be measured by halimeter .

Measurements and time frame: Initial measurements (T0), after two weeks (T1), and after four weeks (T2) ( according to previous studies that uses the same period of time for measurements),17, 18 plaque index (PI), gingival bleeding index (GBI), bracket index and halimeter reading .

During the first week after the start of the study (T0)

ELIGIBILITY:
Inclusion Criteria:

1. participants with fixed orthodontic appliance.
2. participants age 14 years and above and didn't have mental of physical disabilities.
3. participants willing to comply with given oral hygiene instructions.

Exclusion Criteria:

1. patients with mental retardation.
2. patients with systematic diseases.

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-13 (Actual); Primary Completion 2019-06-06 (Estimated); Study Completion 2019-10-11 (Estimated)

PRIMARY OUTCOMES:
Change in volatile sulphur compounds causing halitosis at four weeks. | At baseline then and after four weeks then
  Tanita Breath Checker HC-312SF Fitscan to measures volatile sulphur compounds with six levels of odor.
Change in volatile sulphur compounds causing halitosis at eight weeks. | At four weeks from baseline and after eight weeks then
  Tanita Breath Checker HC-312SF Fitscan to measures volatile sulphur compounds with six levels of odor.

CONTACTS AND LOCATIONS:
Locations (1):
- Riyadh Elm University, Riyadh, Riyadh Region, Saudi Arabia